CLINICAL TRIAL: NCT00124787
Title: A Randomized Double-blind Trial Comparing the Effect of Oral Dimenhydrinate Versus Placebo in Children With Moderate Vomiting Due to Acute Gastroenteritis
Brief Title: A Trial Comparing the Effect of Oral Dimenhydrinate Versus Placebo in Children With Gastroenteritis
Acronym: GAG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Collaborators: Canadian Association of Emergency Physicians (Industry)
Responsible Party: Principal Investigator, Serge Gouin, Associate professor, St. Justine's Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PROJET 2078
Record Dates: First submitted 2005-07-26; First posted 2005-07-28 (Estimated); Last update posted 2012-03-01 (Estimated); Status verified 2012-02

CONDITIONS: Gastroenteritis
MeSH Terms: conditions — Gastroenteritis | interventions — Dimenhydrinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dimenhydrinate (Experimental): dimenhydrinate PO x 4 doses
  Interventions: Drug: Dimenhydrinate
- Placebo (Placebo Comparator): placebo PO x 4 doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dimenhydrinate — Dimenhydrinate PO q 6 hours x 4 doses
  Arms: Dimenhydrinate
Drug: Placebo — Placebo PO q 6 hours x 4 doses
  Arms: Placebo

SUMMARY:
Dimenhydrinate, an over-the-counter, widely used drug in Canada, is an ethanolamine-derivative anti-histamine. It limits the stimulation of the vomiting center by the vestibular system, which is rich in histamine receptors. Multiple studies have shown its effectiveness in treatment of post-operative nausea and vomiting in children. It is also used for treatment of vertigo in children. Furthermore, it has the potential to be much more cost-effective than ondansetron, with an average cost of $0.90 US per dose . Its principal side effects are drowsiness, dizziness and anticholinergic symptoms. Restlessness and insomnia have also been described in children. To date, there has been no published data on the efficacy of dimenhydrinate in controlling emesis in children with acute gastroenteritis.

RESEARCH QUESTION

Do children treated with oral dimenhydrinate during acute gastro-enteritis experience less vomiting episodes than children treated with placebo?

DETAILED DESCRIPTION:
STRUCTURED RESEARCH ABSTRACT

Background: The use of antiemetic drugs to treat nausea and vomiting during an episode of acute gastroenteritis in children remains controversial. To date, there have been a limited number of clinical trials studying this subject matter and health authorities' recommendations are only based on expert opinion. Surveys have shown that despite this lack of evidence, physicians do quite frequently prescribe these drugs. Dimenhydrinate, a histamine receptor blocker, has been proven safe and effective in controlling post-operative nausea and vomiting in children. To our knowledge, no clinical trial has been conducted to study its efficacy in children with acute gastroenteritis.

Objective: To evaluate the efficacy and safety of oral dimenhydrinate in the treatment of vomiting due to acute gastroenteritis in children.

Design: Randomized, double-blind, placebo controlled clinical trial.

Setting: Emergency Department (ED) of an urban pediatric university-affiliated center.

Study population: Children from 1 to 12 years of age presenting to the ED with at least 5 episodes of vomiting in the previous 12 hours and diagnosed with acute gastroenteritis by attending physicians.

Interventions: Study participants will be randomly allocated to receive 8 doses of dimenhydrinate or placebo every six hours (1mg/kg/dose, max dose 50mg/dose)

Primary outcome measure: Number of good outcome, defined as 1 episode or less of vomiting 24 hours after the first dose of drug administration.

Secondary outcome measures: Need for intravenous fluid administration, number and duration of vomiting and diarrhea, side effects, revisit rates and parental absenteeism from work will be compared between the two groups

Sample size and statistics: Based on previously reported data, the researchers estimate that approximately 70% of patients will be free of emesis in the initial 24 hours post medication first dose. The researchers would like to obtain a good outcome in more than 85% with the active medication. With an alpha error of 0.05 and a power of 90%, approximately 90 patients per group will be needed. Patients' characteristics and outcomes will be compared using the Mann Whitney U test and the Chi-square test for categorical variables and the Student's T test for continuous variables. Survival curves will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Children aged from 1 to 12 years old with more than 5 episodes of vomiting in the 12 hours preceding their diagnosis of acute gastroenteritis by an ED attending physician

Exclusion Criteria:

* Pre-existing chronic medical condition such as gastro-intestinal disease, malignancy, metabolic, cardiac, endocrine, immunologic or neurologic disorder
* Suspected secondary diagnosis of surgical abdomen or gynecologic condition, urinary tract infection, migraine or meningitis
* Use of antiemetic therapy within 48 hours prior to ED visit
* Use of medication other than acetaminophen or ibuprofen in the previous 48 hours
* History of allergy or adverse reaction to dimenhydrinate
* Severe dehydration requiring immediate intravenous fluid therapy
* Hematemesis or hematochezia

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2005-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Number of good outcome, defined as 1 episode or less of vomiting 24 hours after the first dose of drug administration. | 24 hours

SECONDARY OUTCOMES:
Need for intravenous fluid administration | 24 hours
Number and duration of vomiting and diarrhea | 7 days
Side effects | 7 days
Revisit rates | 7 days
Parental absenteeism from work will be compared between the two groups | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Serge Gouin, MDCM, FRCPC, Principal Investigator — Ste-Justine Hospital, Department of Pediatrics, Montreal University
Locations (1):
- Ste-Justine Hospital, Montreal, Quebec, Canada